CLINICAL TRIAL: NCT02878746
Title: Robotic Mirror Therapy System for Functional Recovery of Hemiplegic Arms
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Collaborators: Seoul National University (Other)
Responsible Party: Principal Investigator, Sun Gun Chung, Professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SNUH-1209-051-425
Record Dates: First submitted 2016-08-15; First posted 2016-08-25 (Estimated); Last update posted 2021-04-02 (Actual); Status verified 2021-03

CONDITIONS: Stroke
Keywords: Mirror therapy; Proprioception; Rehabilitation; Stroke; Hemiplegia
MeSH Terms: conditions — Stroke; Hemiplegia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Robotic mirror therapy (Experimental): For 30 min per day for two weeks (10 sessions)
  Interventions: Device: Robotic mirror therapy
- Conventional mirror therapy (Active Comparator): For 30 min per day for two weeks (10 sessions)
  Interventions: Device: Conventional mirror therapy

INTERVENTIONS:
Device: Robotic mirror therapy — 2-dimensional
  Arms: Robotic mirror therapy
Device: Conventional mirror therapy — 2- and 3-dimensional
  Arms: Conventional mirror therapy

SUMMARY:
The investigators developed a real-time 2-axis mirror robot system as a simple add-on module for conventional mirror therapy using a closed feedback mechanism, which allows for real-time movement of the hemiplegic arm. The investigators conduct a case study for stroke patients with a two-dimensional mirror robot for 30 min per day for two weeks (10 sessions). For the conventional mirror therapy group, the investigators prepared the tasks for fine motor training.

DETAILED DESCRIPTION:
The investigators conduct a case study for stroke patients with a two-dimensional mirror robot for 30 min per day for two weeks (10 sessions). For the conventional mirror therapy group, the investigators prepared the tasks for fine motor training. These tasks included more complicated tasks so that the participants would be interested in the tasks without the robot system.

Before and after 10 sessions of the therapy, the investigators conduct functional evaluations: the Fugl-Meyer assessment scale of the upper extremity (FMA-UE), the modified Ashworth scale, the modified Barthel index of upper extremity (MBI-UE: personal hygiene, bathing, feeding, and dressing), and the Jebsen hand function test, hand power measurement, and hemispatial neglect test (line bisection test and Albert's test) with the same occupational therapist. The motor evoked potential was measured for the patients without the history of brain surgery or seizure.

The investigators selected a thumb finding test (TFT) among various tools for assessing proprioception, because TFT is widely used and reliable. The TFT can be assessed, after confirming normal proprioception in the unaffected arm, by the patient touching the nose with their eyes closed while the examiner lifts the affected arm to eye level. The patient is then asked to grasp the thumb of the affected hand with the unaffected hand, and this is repeated. The examiner then places a hand over the patient's eyes and raises the patient's affected hand to well above the patient's head. The patient is then asked to grasp the thumb as before.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years old
* Supratentorial stroke diagnosed between 4 months and 6 years ago
* Upper-limb hemiplegia with Medical Research Council grade 2 or less.

Exclusion Criteria:

* Severe spasticity with modified Ashworth scale of grade 3 or more;
* Mini-mental state examination score less than 12
* Global or sensory aphasia.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Fugl-Meyer assessment scale | Change from baseline data at 2 weeks

SECONDARY OUTCOMES:
Thumb finding test | Before treatment, after 2 weeks, after 2 months
Modified Ashworth scale | Before treatment, after 2 weeks, after 2 months
Modified Barthel index | Before treatment, after 2 weeks, after 2 months
Hand power(lb) assessed by dynamometer | Before treatment, after 2 weeks, after 2 months
Jebsen hand function test | Before treatment, after 2 weeks, after 2 months
Hemispatial neglect test | Before treatment, after 2 weeks, after 2 months
Functional brain MRI | Before treatment, after 2 weeks
Fugl-Meyer assessment scale | after 2 months

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hamzei F, Lappchen CH, Glauche V, Mader I, Rijntjes M, Weiller C. Functional plasticity induced by mirror training: the mirror as the element connecting both hands to one hemisphere. Neurorehabil Neural Repair. 2012 Jun;26(5):484-96. doi: 10.1177/1545968311427917. Epub 2012 Jan 13. PMID 22247501
- [Background] Pandian JD, Arora R, Kaur P, Sharma D, Vishwambaran DK, Arima H. Mirror therapy in unilateral neglect after stroke (MUST trial): a randomized controlled trial. Neurology. 2014 Sep 9;83(11):1012-7. doi: 10.1212/WNL.0000000000000773. Epub 2014 Aug 8. PMID 25107877
- [Background] Dohle C, Pullen J, Nakaten A, Kust J, Rietz C, Karbe H. Mirror therapy promotes recovery from severe hemiparesis: a randomized controlled trial. Neurorehabil Neural Repair. 2009 Mar-Apr;23(3):209-17. doi: 10.1177/1545968308324786. Epub 2008 Dec 12. PMID 19074686
- [Background] Thieme H, Bayn M, Wurg M, Zange C, Pohl M, Behrens J. Mirror therapy for patients with severe arm paresis after stroke--a randomized controlled trial. Clin Rehabil. 2013 Apr;27(4):314-24. doi: 10.1177/0269215512455651. Epub 2012 Sep 7. PMID 22960240
- [Background] Bhasin A, Padma Srivastava MV, Kumaran SS, Bhatia R, Mohanty S. Neural interface of mirror therapy in chronic stroke patients: a functional magnetic resonance imaging study. Neurol India. 2012 Nov-Dec;60(6):570-6. doi: 10.4103/0028-3886.105188. PMID 23287316